CLINICAL TRIAL: NCT05989841
Title: Mitigating PTSD-CUD Among Women Presenting to Emergency Care After Sexual Assault: Testing a Digital Therapeutic Targeting Anxiety Sensitivity
Brief Title: Mitigating PTSD-CUD After Sexual Assault
Acronym: RISE-C
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); National Institute on Drug Abuse (NIDA) (NIH); Hennepin HART (Unknown); Tulsa Police Department Forensic Nursing (Unknown); SAFE Austin Harbor Shelter (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UNLV-2023-649; 1K23DA054299-01 (NIH)
Record Dates: First submitted 2023-05-10; First posted 2023-08-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Posttraumatic Stress Disorder; Cannabis Use Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RISE Guide (Experimental): Brief cognitive behavioral intervention completed in the 3 weeks post-assault delivered via Internet on participants' smartphones targeting anxiety sensitivity, or fear of anxious arousal. Patients learn psychoeducation regarding the nature of stress, cognitive retraining to reduce negative interpretations of stress, and how to complete interoceptive exposures to reduce anxiety sensitivity. These skills are supported by 6 concurrent then subsequent weeks of ecological momentary intervention to deliver personalized intervention reminders based on symptoms.
  Interventions: Behavioral: RISE Guide
- Relaxation (Active Comparator): Patients will download the "Breathe2Relax" app, which delivers information about how to use diaphragm breathing (taking slow, deep breaths through the diaphragm) to manage stress. Participants will receive reminders to engage with the intervention. Participants will also receive ecological momentary intervention reminders to engage with the relaxation intervention.
  Interventions: Behavioral: Relaxation Control

INTERVENTIONS:
Behavioral: RISE Guide — Brief cognitive behavioral intervention completed in the 3 weeks post-assault delivered via Internet on participants' smartphones targeting anxiety sensitivity, or fear of anxious arousal. Patients learn psychoeducation regarding the nature of stress, cognitive retraining to reduce negative interpretations of stress, and how to complete interoceptive exposures to reduce anxiety sensitivity. These skills are supported by 6 concurrent then subsequent weeks of ecological momentary intervention to deliver personalized intervention reminders based on symptoms.
  Arms: RISE Guide
Behavioral: Relaxation Control — Patients will download the "Breathe2Relax" app, which delivers information about how to use diaphragm breathing (taking slow, deep breaths through the diaphragm) to manage stress. Participants will receive reminders to engage with the intervention. Participants will also receive ecological momentary intervention reminders to engage with the relaxation intervention.
  Arms: Relaxation

SUMMARY:
683,000 women are sexually assaulted annually in the United States, half of whom develop chronic posttraumatic stress disorder (PTSD) and thus have markedly increased risk for cannabis use disorder (CUD). The current proposal will test the acceptability, initial efficacy, and mechanisms underlying a novel digital therapeutic targeting risk for PTSD-CUD, which could address the critical need for PTSD-CUD prevention for the 100,000 women who annually present for emergency care after sexual assault. In this research context, the applicant will receive key training in multisite, emergency-care based randomized clinical trials (RCTs), advanced statistical analyses for RCTs and ecological momentary assessment data, biobehavioral mechanisms underlying PTSD-CUD prevention, and professional development, launching her independent research career focused on reducing the public health burden of PTSD-CUD among sexual assault survivors by leveraging digital therapeutics.

ELIGIBILITY:
Inclusion Criteria:

1. Women sexual assault survivors presenting for emergency care <72 hours post-assault at 1 of our 4 emergency care sites
2. English speakers
3. 18+ years of age
4. Able to provide informed consent
5. Have a smartphone with continuous service >1 year
6. Report >1x/weekly cannabis use on a substance use screener
7. Report elevated AS (>17 on the Anxiety Sensitivity Index-3)

Exclusion Criteria:

1. Inability to provide informed consent (e.g., serious injury preventing the ability to hear, speak, or see to consent and participate, or other causes (e.g., diagnosed cognitive deficits, diagnosed dementia, asleep at time of screening)).
2. Prisoner
3. Currently pregnant
4. Lives with assailant and plans to continue to do so
5. Admitted patient
6. No mailing address
7. Previously enrolled
8. No sexual assault nurse examiner (SANE) examination
9. Reporting current plan and intent for suicide or homicide
10. Does not understand written and spoken English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Assigned female at birth and currently identifying as female
Enrollment: 68 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Anxiety Sensitivity Index-3 (ASI-3) | 6 weeks
  18-item self-report measure of anxiety sensitivity assessing all three subdomains of anxiety sensitivity (physical, cognitive, social). Participants respond to 18 items (e.g., It scares me when my heart beats rapidly) on a 4-point Likert scale. Scores range from 0-72, with higher scores indicating higher levels of anxiety sensitivity.

SECONDARY OUTCOMES:
Marijuana Problems Scale (MPS) | 6 months
  19-item self-report measure of problems related to cannabis use (e.g., problems with work, school, social functioning). Participants rate 19 items on a 3- point Likert scale. Scores range from 0 to 38, with higher scores indicating more problems related to cannabis use.
Marijuana Motives Measure - Coping | 6 months
  The MMM is a 25-item self-report measure of cannabis motives, including coping-oriented motives for cannabis use. Participants respond to a list of motives (e.g., to forget my worries, to get high) on a 5-point Likert scale. Scores range from 25 to 125 for the entire measure, with higher scores indicating higher levels of various types of marijuana motives. The primary motive that will be used as an outcome is coping motives (scores range from 4 to 20 on this subscale).
Patient Reported Outcome Measurement Information System - Anxiety Measurement Information System (PROMIS) Anxiety and Depression | 6 months
  7-items assessing self-reported symptoms of anxiety (e.g., anxious, worried, nervous) rated on a 5-point scale. Scores range from 7 to 35, with higher scores indicating higher levels of anxiety. T-scores are used for final scoring.
Patient Reported Outcome Measurement Information System - Depression Measurement Information System (PROMIS) Anxiety and Depression | 6 months
  8 items assessing self-reported symptoms of depression (e.g., worthlessness, helplessness, sadness) rated on a 5-point scale. Scores range from 8 to 40, with higher scores indicating higher levels of depression. T-scores are used for final scoring.
Cannabis Use Frequency | 6 weeks
  Ecological momentary assessment will include self-report measures of whether or not cannabis was used that day (yes/no). The item will be scored as 0 (no) vs. 1 (yes), with higher scores indicating higher levels of cannabis use frequency.
Cannabis Use Quantity | 6 weeks
  Ecological momentary assessment will assess quantity of cannabis used on an 8-point scale, assessed 1x/day over 6 weeks. Scores will range from 1-8, with higher scores indicating a higher quantity of cannabis consumed.
Marijuana Cravings - Emotionality Questionnaire | 6 weeks
  Ecological momentary assessment will include a state version of the emotionality subscale of the Marijuana Cravings Questionnaire. This consists of 4 items rated on a 7-point Likert scale, assessed 4x/day over 6 weeks. Scores range from 4 to 28, with higher scores indicating higher levels of cravings.
PTSD Checklist for Diagnostic and Statistical Manual -5 (DSM-5) (PCL-5) | 6 months
  20-item self-report measure of DSM-5 PTSD symptoms, including 4 symptom clusters of PTSD (re-experiencing, avoidance, negative alterations in cognition and mood, alterations in arousal and reactivity). Participants respond to items corresponding to each DSM-5 symptom of PTSD on a 5-point Likert scale (0 to 4). Scores range from 0 to 80, with higher scores indicating higher levels of PTSD symptoms.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Hennepin Assault Response Team, Minneapolis, Minnesota
  - University Medical Center, Las Vegas, Nevada
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Harbor Shelter, Smithfield, North Carolina
  - Tulsa Forensic Nursing, Tulsa, Oklahoma
  - SAFE Austin, Austin, Texas